CLINICAL TRIAL: NCT03162510
Title: An Phase I Dose-Escalation Study of Biweekly Abraxane in Combination With Oxaliplatin and Oral S-1/LV (SOLAR Regimen) as First-line Chemotherapy in Patients With Advanced Gastric, Pancreatic and Biliary Cancers
Brief Title: Biweekly SOLAR, as First-line C/T in Pts With Gastric, Pancreatic and Biliary Cancers
Acronym: SOLAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Cheng-Kung University Hospital (Other); National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCOG T1216
Record Dates: First submitted 2016-11-15; First posted 2017-05-22 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2021-06

CONDITIONS: Gastric Cancer in Situ; Pancreatic Cancers; Biliary Cancers
Keywords: SOLAR regimen
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms | interventions — Oxaliplatin; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; S 1 (combination); Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SOLAR (Experimental): Albumin-Bound Paclitaxel /nab-Paclitaxel (Abraxane®) 150 mg/m2 IVD 30 min followed by Oxaliplatin 60~ 85 mg/m2 IVD 2hr at D1, plus Tegafur,oral S-1 35mg/m2 and Folinic acid/LV 30mg twice daily from D1 to D7, every 14 days as a cycle till disease progression
  Interventions: Drug: Oxaliplatin; Drug: Albumin-Bound Paclitaxel /nab-Paclitaxel; Drug: S-1; Drug: LV

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin 60 - 85 mg/m2 IVD 2hr at D1, every 14 days as a cycle till disease progression
  Other Names: Oxalip
Drug: Albumin-Bound Paclitaxel /nab-Paclitaxel — 150 mg/m2 IVD 30 min bi-weekly.
  Other Names: Abraxane
Drug: S-1 — Tegafur,oral S-1 35mg/m2 twice daily from D1 to D7, every 14 days as a cycle till disease progression.
  Other Names: Tegafur,
Drug: LV — LV 30mg twice daily from D1 to D7, every 14 days as a cycle till disease progression
  Other Names: Lecovorin

SUMMARY:
The primary purpose of the study is to determine the maximal tolerated dose (MTD) of Oxaliplatin in this phase I study. The secondary objectives are to determine the response rate, progression free survival, overall survival, and safety profiles.

Eligible patients will receive a triplet chemotherapy consisting of nab-paclitaxel (Abraxane®) 150 mg/m2 IVD 30 min followed by Oxaliplatin 60 - 85 mg/m2 IVD 2hr at D1, plus oral S-1 35mg/m2 and Leucovorin 30mg twice daily from D1 to D7, every 14 days as a cycle till disease progression.

DETAILED DESCRIPTION:
Eligible patients will receive a triplet chemotherapy consisting of nab-paclitaxel (Abraxane®) 150 mg/m2 IVD 30 min followed by Oxaliplatin 60 - 85 mg/m2 IVD 2hr at D1, plus oral S-1 35mg/m2 and Leucovorin 30mg twice daily from D1 to D7, every 14 days as a cycle till disease progression.

In this study (a standard 3 x 3 design), patients will be enrolled in cohort of 3 to receive escalating dose of Oxaliplatin at three dose levels (level I, 60 mg/m2, level II, 75 mg/m2 and level III, 85 mg/m2). Intra-patient dose escalation will not be allowed. If none of the first 3 patients of a cohort experiences a dose limiting toxicity (DLT), then dose escalation will proceed for next cohort of patients. If 1 of 3 patients developed DLT, the cohort will be expanded to 6 patients. If ≤2 patients of the 6 patients experience DLT, then dose escalation will proceed in next study cohort unless 85 mg/m2 have reached. If 2 of the first 3 or ≥3 of 6 patients developed DLT at certain dose level, then dose escalation will be withheld and the prior dose level will be the maximum tolerated dose (MTD). A minimum of 6 evaluable patients will be treated at the MTD dose level with no more than 2 of the 6 patients having DLT at this dose level. The MTD will be considered as the recommended dose for future Phase II studies. The number of patient accrual will range from 12 and 18 (6/dose level) evaluable patients in the dose-finding stage to determine the MTD of Oxaliplatin in this combination regimen.

Of patients who experience grade 2 sensory neuropathy after the triplet chemotherapy, Oxaliplatin will be omitted (only nab-paclitaxel plus S-1/LV will be continued) until the recovery of sensory neuropathy to grade 1 or less then Oxaliplatin will be re-instituted.

CBC/DC, AST/ALT and BUN/Cr will be determined at baseline and every 2 weeks during study period. Serum level of albumin, bilirubin (T), LDH, Alk-P/GGT, Na/K/Mg/Ca/P and CRP will be determined at baseline and every 4 weeks during the treatment. Radiographic objective tumor response assessment, according to RECIST version 1.1, by CT scan or MRI at baseline, and then every 6 weeks during the study period. Tumor marker, CEA and CA 19-9, will be evaluated at baseline and every 4 weeks during the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma or carcinoma of the stomach, pancreas and biliary tract with unresectable, recurrence or metastatic disease.
* No prior systemic chemotherapy except adjuvant chemotherapy that has completed 6 months prior enrollment.
* Palliative RT to bone but not the primary, main tumor site is permitted.
* At least one measurable lesion over non-radiated site.
* Aged between 20 to 70 years old.
* ECOG Performance Status <= 1.
* Life expectancy greater than 12 weeks.
* Adequate bone marrow function : absolutely neutrophil count >= 1.5 x 109/L or WBC >= 4 x 109/L, hemoglobin >= 9 g/dl, platelet count 100 x 109/L
* Adequate liver function : ALT <= 2.5 x ULN and Bilirubin < 1.5 x ULN
* Adequate renal function: creatinine < 1.5 x ULN and calculated eGFR> 50 mL/min.

Exclusion Criteria:

* Major surgery within four weeks prior to study enrolment.
* Patient with Ampulla vater cancer is excluded.
* Patients with suspicious or history of CNS metastasis.
* Patients who with active or uncontrolled infections.
* Patients who have history of myocardial infarction or unstable angina within 6 months before entry.
* Patients with concomitant illness that might be aggravated by chemotherapy.
* Patients who are pregnant or with breast feeding.
* Other concomitant or previously malignancy within 3 yrs except for in situ cervix cancer or squamous cell carcinoma of the skin, stage 0-I colon or breast treated by surgery only and without evidence of relapsed tumor.
* Mental status is not fit for clinical trial
* Fertile men and women unless using a reliable and appropriate contraceptive method.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
MTD of Oxaliplatin | From date of registration until the date of definition of MTD or first documented progression or date of death from any cause, whichever came first, assessed up to 28weeks.
  Dose-limiting toxicity (DLT),patients will be enrolled in cohort of 3 to receive escalating dose of Oxaliplatin at three dose levels (level I, 60 mg/m2, level II, 75 mg/m2 and level III, 85 mg/m2)or more of defined events.

SECONDARY OUTCOMES:
tumor response | From date of registration until the date of definition of MTD or first documented progression or date of death from any cause, whichever came first, assessed up to 28weeks.
  Efficacy evaluations: objective tumor response according to RECIST 1.1
Overall survival | Overall survival will be assessed. From date of registration until the date of death, assessed up to 60 months.
  Overall survival: defined as the time from the date of first study treatment to the date of patient death, due to any cause, or to the last date the patient was known to be alive. The primary analysis population for the overall survival will be per-protocol population. The endpoint will also be analyzed in the intent-to-treat population. Kaplan-Meier estimates will be calculated for the overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, MD PHD, Study Chair — National Health Research Institutes, Taiwan
Locations (1):
- Taiwan Cooperative Oncology Group, National Health Research Institutes, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsai HJ, Yang SH, Hsiao CF, Kao HF, Su YY, Shan YS, Yen CJ, Du JS, Hsu C, Wu IC, Chen LT. A phase 1 study of biweekly nab-paclitaxel/oxaliplatin/S-1/LV for advanced upper gastrointestinal cancers: TCOG T1216 study. Oncologist. 2024 Oct 3;29(10):e1396-e1405. doi: 10.1093/oncolo/oyae109. PMID 38902994